CLINICAL TRIAL: NCT02265497
Title: Brazilian Network for Lymphoma Registry
Acronym: Relinfo
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Claudio Gustavo Stefanoff (Other Government)
Collaborators: Adriana Alves de Souza Scheliga (Unknown); Claudete Esteves Nogueira Pinto Klumb (Unknown); Ricardo de Sá Bigni (Unknown); Luciana Wernersbach Pinto (Unknown); Rocio Hassan (Unknown); Isabele Avila Small (Unknown); Monik Mariano Pinto (Unknown); Cecilia Ferreira da Silva (Unknown)
Responsible Party: Sponsor-Investigator, Claudio Gustavo Stefanoff, Claudio Gustavo Stefanoff, Instituto Nacional de Cancer, Brazil
Organization: Instituto Nacional de Cancer, Brazil (Other Government)
Other Study IDs: Relinfo
Record Dates: First submitted 2014-09-18; First posted 2014-10-16 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2016-08

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hodgkin's or non-Hodgkin lymphoma: All patients with diagnoses of Hodgkin's or non-Hodgkin lymphoma with available with available clinical, histopathology and treatment data.

SUMMARY:
Currently there are no official data concerning incidence, progression and prognosis of patients with lymphoma in Brazil.This project aims the establishment of a network of 12 Brazilian Institutions to implement a Lymphoma Registry (RELINFO) with the Brazilian National Cancer Institute (INCA) as the Coordinating Center.We intend to develop and implement a computerized system for data entry and information management of patients with lymphomas. This will enable create a virtual registry of demographic, clinical, epidemiological, histopathological, molecular, and therapeutic data. This clinical record must be linked to histopathological and molecular diagnosis, allowing institutions that work in the context of the public health system have access to new technologies for early cancer diagnosis.We expect is that this record reliably portrays the scene of lymphomas in our state and will become a management model that can be replicated at the national level. Thus, the implementation of RELINFO will strengthen the multidisciplinary diagnosis, promote the standardization of clinical record of patients with lymphomas and provide subsidies to cooperative research projects between participating institutions.

DETAILED DESCRIPTION:
Data collection and management:

For data collection will use a common system for all institutions participating.We developed a computerized tool that utilizes models of case report forms (CRF) and allows the inclusion and management of clinical, epidemiological, histopathological and molecular data. The clinical and laboratory data of patients included in RELINFO will be obtained from the hospital records. The integration of local databases allows constitute the RELINFO, conceived as a virtual database of patients with lymphoma. The INCA as Coordinating Center is committed to the security of this database.Standardization of diagnosisThis phase includes structuring a technological platform for the standardization of histopathologic diagnosis (establishing common routines in hematopathology) and the incorporation of molecular methods in the diagnosis of lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* All patients (adult or child) with diagnosis of Hodgkin's or non-Hodgkin lymphoma with available with available clinical, histopathology and treatment data
* Patient enrolled on study sites included on this project

Exclusion Criteria:

* Patients (adult or child) with other diagnoses of cancer

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with diagnosis of Hodgkin's or non-Hodgkin lymphoma with available with available clinical, histopathology and treatment data.
Sampling Method: Non-Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2014-03; Primary Completion 2018-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
rate of incidence of lymphomas in Brazil | 6 years
  Identify the current situation of lymphomas, through the deployment of a Lymphoma Registry in cancer treatment centers of Rio de Janeiro, Brazil

SECONDARY OUTCOMES:
epidemiological characterization of lymphomas in Brazil | 6 years
  description of demographic, clinical, epidemiological, histopathological, molecular, and therapeutic data of lymphoma patients
establishing common routines in hematopathology | 6 years
  Structure a technology platform that allows the standardization of histopathological diagnosis and the incorporation of molecular methods in the diagnosis of lymphoma.

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Gustavo Stefanoff, Doctor, Study Director — Instituto Nacional de Cancer, Brazil
Locations (1):
- Brazilian National Cancer Institute - INCA/ Ministry Of HealthClinical Research Department, Rio de Janeiro, Rio de Janeiro, Brazil